CLINICAL TRIAL: NCT07124585
Title: Short-Term Effect of Non-Nutritive Sweeteners (Sucralose and Saccharin) Consumption on Glycaemic Control and Gut Microbiota in Type 2 Diabetes Patients
Brief Title: Short-Term Effects of Sucralose and Saccharin on Blood Sugar and Gut Microbiota in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Monash University Malaysia (Other)
Responsible Party: Principal Investigator, Harvinder Kaur A/P Gilcharan Singh, Lecturer, National University of Malaysia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FRGS/1/2024/SKK06/UKM/03/4
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Non-nutritive sweetener; artificial sweetener; gut microbiota; saccharin; sucralose; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trichlorosucrose; Saccharin; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crossover Arm 1 (Sucralose) (Active Comparator): Each participant will receive all three interventions, sucralose, saccharin, and placebo in a randomized sequence over three separate phases. Each intervention phase lasts for seven consecutive days and is separated by a washout period of 4 weeks to minimize carryover effects.
  Interventions: Dietary Supplement: Sucralose
- Crossover Arm 2 (Saccharin) (Active Comparator): Each participant will receive all three interventions, sucralose, saccharin, and placebo in a randomized sequence over three separate phases. Each intervention phase lasts for seven consecutive days and is separated by a washout period of 4 weeks to minimize carryover effects.
  Interventions: Dietary Supplement: Saccharin
- Crossover Arm 3 (Placebo) (Placebo Comparator): Each participant will receive all three interventions, sucralose, saccharin, and placebo in a randomized sequence over three separate phases. Each intervention phase lasts for seven consecutive days and is separated by a washout period of 4 weeks to minimize carryover effects.
  Interventions: Other: Placebo (Calcium Carbonate)

INTERVENTIONS:
Dietary Supplement: Sucralose — Participants will consume one capsule containing sucralose 5mg/kg body weight, with the dosage individualized according to body weight. The capsule will be taken once daily in the morning, after breakfast, with plain water. This intervention will last for seven consecutive days.
  Arms: Crossover Arm 1 (Sucralose)
Dietary Supplement: Saccharin — Participants will consume one capsule containing saccharin 2mg/kg body weight, with the dosage individualized according to body weight. The capsule will be taken once daily in the morning, after breakfast, with plain water. This intervention will last for seven consecutive days.
  Arms: Crossover Arm 2 (Saccharin)
Other: Placebo (Calcium Carbonate) — Participants will consume one capsule per day, containing a fixed dose of 500 mg. The capsule will be taken once daily in the morning, after breakfast, with plain water. This intervention will last for seven consecutive days.
  Arms: Crossover Arm 3 (Placebo)

SUMMARY:
This clinical trial investigates the short-term effects of two commonly used non-nutritive sweeteners (NNS), saccharin and sucralose, on blood glucose regulation and the gut microbiota in adults with Type 2 Diabetes Mellitus (T2DM). While NNS are widely promoted as sugar substitutes to aid glycaemic control, emerging evidence suggests that even small doses may influence metabolic health, potentially through interactions with the gut microbial community.

The study is designed as a double-blind, randomized, placebo-controlled, crossover trial involving 33 adults with T2DM. Each participant will receive all three interventions, saccharin, sucralose, and a placebo (calcium carbonate) in random order. Each intervention will be administered once daily in capsule form for 7 consecutive days, with a 4-week washout period between phases to minimize carryover effects.

Throughout the trial, data will be collected on anthropometry, blood-based glycaemic biomarkers, dietary intake, physical activity, and stool samples. Gut microbiota composition will be assessed via 16S rRNA gene sequencing.

The primary aim is to generate evidence on whether short-term exposure to NNS can affect glycaemic outcomes and gut microbial profiles in individuals with T2DM. The findings are expected to support future dietary recommendations on NNS use and improve our understanding of diet-microbiota-host interactions, particularly within Asian populations.

DETAILED DESCRIPTION:
Although these sweeteners are generally recognized as safe, emerging studies have raised concerns regarding their potential metabolic effects. In particular, findings on their influence on glycaemic control in humans remain inconsistent. One proposed mechanism underlying these effects involves modulation of the gut microbiota, which is increasingly recognised as a critical regulator of host metabolic homeostasis. However, current evidence in human studies is limited and inconclusive.

Individuals with T2DM commonly exhibit pre-existing gut dysbiosis, raising important questions about whether the use of NNS may further impair microbial composition or function. To date, no clinical trial has comprehensively examined the short-term effects of sucralose and saccharin on both glycaemic responses and the gut microbiota in specific T2DM population. Moreover, data from Asian populations whose dietary patterns, gut microbial composition, and metabolic phenotypes differ significantly from Western cohorts are scarce. Given the widespread consumption of NNS in daily diets, especially among individuals seeking glycaemic control, this represents a critical evidence gap with potential implications for dietary recommendations and metabolic health.

This study aims to address these gaps through a clinical trial in adults with T2DM. The crossover design enables within-subject comparisons, thereby reducing inter-individual variability and enhancing statistical power to detect subtle biological effects. Reference to previous studies has shown inconsistencies arising from factors such as inconsistent dosing, varying administration routes (e.g., sachet vs. capsule; pure compound vs. commercial product), differences in intervention duration, and a lack of control for confounding variables such as habitual diet, medication use, and physical activity. To address these issues, we have incorporated several methodological improvements. Our study will implement a body weight-based individual dosing protocol, oral administration in a standardised pure compound capsule form, and detailed characterisation of participants' dietary intake and lifestyle behaviours.

Additionally, for our study phenotype, we have strictly controlled for patients' diabetes progression, including diagnosis duration (1-5 years), treatment type (oral antidiabetic medication only, no insulin), age group (30-50 years), demographic (male only), ethnicity (single ethnic group), and BMI range (specified). Through these measures, our study aims to minimise variability, particularly in gut microbiota outcomes and generate more robust results.

ELIGIBILITY:
Inclusion criteria This study aims to recruit a cohort of patients with early-phase diagnosed T2DM whose conditions are stable that can best represent the Malaysian DM phenotypes.

1. Male citizens of Malaysia.
2. Aged between 30 and 59 years.
3. BMI between 23-29.9 kg/m² (Overweight).
4. Diagnosed with diabetes for a duration between 1-10 years.
5. Currently on oral antidiabetic medications and not on insulin.
6. Initial HbA1c less than 10%.
7. Patients with other stable, non-severe chronic conditions (e.g., hypertension, dyslipidemia) may be included if they have been on a stable prescribed oral treatment for at least 6 months.
8. Patients who have undergone dietary counselling for diabetes and are willing to maintain their habitual diabetes-friendly diet and usual physical activity patterns throughout the study period.
9. Willing to refrain from alcohol throughout the study period.
10. Must be literate in English or Bahasa Malaysia.

Exclusion criteria The exclusion criteria will primarily focus on lifestyle behaviours or dietary practices that deviate from typical Malaysian lifestyles and while also considering behaviours that could significantly alter the gut microbiota.

1. Current smoking, alcohol use, or drug abuse.
2. Experienced more than a 5% change in body weight within the past 3 months.
3. Acute illness or significant cardiovascular, psychological, neurological, renal, or endocrine diseases, apart from diabetes.
4. Intolerance or allergy to test products.
5. Special dietary practices (e.g., intermittent fasting, vegetarian, ketogenic diet) that deviate from typical Malaysian dietary patterns.
6. Treatment with glucocorticoids, antibiotics or other medications and food supplements (e.g. probiotics) that can significantly alter intestinal function and gut microbiome.
7. Involvement in clinical trials within the last 3 months.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 33 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control | 6 months
  The primary outcome of this study is to assess the change in glycaemic control, measured by insulin sensitivity using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), which will be calculated from fasting glucose and insulin levels following NNS consumption

SECONDARY OUTCOMES:
Gut microbiota composition and diversity | 6 months
  The secondary outcome is to evaluate changes in gut microbiota composition and diversity following NNS consumption. Microbiota outcomes will be assessed via 16S rRNA gene sequencing. Alpha diversity and beta diversity metrics will be used to evaluate within- and between-group microbiota differences. Differential abundance analysis will be conducted to identify specific taxanomy associated with each intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Kesihatan Setapak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data including glycaemic parameters and gut microbiota profiles.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data (IPD), study protocol, SAP, ICF, and analytic code will be available beginning 6 months after publication of the primary results and will remain available for 5 years thereafter. Extensions may be considered upon request. Data will not be available before publication.
Access Criteria: Access to de-identified IPD and supporting documents will be granted to qualified researchers affiliated with academic institutions or non-profit organizations for scientific purposes only. Requests must include a methodologically sound proposal and be reviewed by the principal investigator and the study's ethics committee. Approved data will be shared through secure institutional data-sharing platforms or encrypted transfer, under a data use agreement that ensures participant confidentiality and responsible data handling.

REFERENCES:
- [Result] Suez J, Korem T, Zeevi D, Zilberman-Schapira G, Thaiss CA, Maza O, Israeli D, Zmora N, Gilad S, Weinberger A, Kuperman Y, Harmelin A, Kolodkin-Gal I, Shapiro H, Halpern Z, Segal E, Elinav E. Artificial sweeteners induce glucose intolerance by altering the gut microbiota. Nature. 2014 Oct 9;514(7521):181-6. doi: 10.1038/nature13793. Epub 2014 Sep 17. PMID 25231862
- [Result] Serrano J, Smith KR, Crouch AL, Sharma V, Yi F, Vargova V, LaMoia TE, Dupont LM, Serna V, Tang F, Gomes-Dias L, Blakeslee JJ, Hatzakis E, Peterson SN, Anderson M, Pratley RE, Kyriazis GA. High-dose saccharin supplementation does not induce gut microbiota changes or glucose intolerance in healthy humans and mice. Microbiome. 2021 Jan 12;9(1):11. doi: 10.1186/s40168-020-00976-w. PMID 33431052
- [Result] Suez J, Cohen Y, Valdes-Mas R, Mor U, Dori-Bachash M, Federici S, Zmora N, Leshem A, Heinemann M, Linevsky R, Zur M, Ben-Zeev Brik R, Bukimer A, Eliyahu-Miller S, Metz A, Fischbein R, Sharov O, Malitsky S, Itkin M, Stettner N, Harmelin A, Shapiro H, Stein-Thoeringer CK, Segal E, Elinav E. Personalized microbiome-driven effects of non-nutritive sweeteners on human glucose tolerance. Cell. 2022 Sep 1;185(18):3307-3328.e19. doi: 10.1016/j.cell.2022.07.016. Epub 2022 Aug 19. PMID 35987213
- [Result] Gryglewski RJ, Swies J, Chlopicki S, Niezabitowski P. Permissive effect of molsidomine towards cardioprotective action of iloprost in myocardial ischemia in cats. J Physiol Pharmacol. 1993 Sep;44(3):313-8. PMID 7694690
- [Result] Frisch SM, Francis H. Disruption of epithelial cell-matrix interactions induces apoptosis. J Cell Biol. 1994 Feb;124(4):619-26. doi: 10.1083/jcb.124.4.619. PMID 8106557
- [Result] Pesak J, Peutelschmiedova A. [Elucidation of the etiology of spastic dysphemia]. Acta Univ Palacki Olomuc Fac Med. 1986;115:7-29. No abstract available. French. PMID 2951976
- [Result] Clark DJ, Tan KS, Lipworth BJ. Evaluation of plasma and urinary salbutamol levels in COPD. Eur J Clin Pharmacol. 1996;51(1):91-3. doi: 10.1007/s002280050166. PMID 8880058
- [Result] Thomson P, Santibanez R, Aguirre C, Galgani JE, Garrido D. Short-term impact of sucralose consumption on the metabolic response and gut microbiome of healthy adults. Br J Nutr. 2019 Oct 28;122(8):856-862. doi: 10.1017/S0007114519001570. Epub 2019 Sep 13. PMID 31258108
- [Result] Zhou Z, Sun B, Yu D, Zhu C. Gut Microbiota: An Important Player in Type 2 Diabetes Mellitus. Front Cell Infect Microbiol. 2022 Feb 15;12:834485. doi: 10.3389/fcimb.2022.834485. eCollection 2022. PMID 35242721
- [Result] Toews I, Lohner S, Kullenberg de Gaudry D, Sommer H, Meerpohl JJ. Association between intake of non-sugar sweeteners and health outcomes: systematic review and meta-analyses of randomised and non-randomised controlled trials and observational studies. BMJ. 2019 Jan 2;364:k4718. doi: 10.1136/bmj.k4718. PMID 30602577
- [Derived] Tan HS, Gilcharan Singh HK, Mariappan V, Jamil NA, Mustapa SN, Misra S. Short-Term Effects of Nonnutritive Sweetener (Sucralose and Saccharin) Consumption on Glycemic Control and Gut Microbiota in Patients With Type 2 Diabetes: Protocol for a Double-Blind, Randomized, Placebo-Controlled, Crossover Trial. JMIR Res Protoc. 2025 Dec 10;14:e82695. doi: 10.2196/82695. PMID 41370820